CLINICAL TRIAL: NCT03860402
Title: The Effect of Warm Local Anesthetic Solution for Sensory Block on Epidural Anesthesia of Cesarean Delivery : a Randomized Controlled Study
Brief Title: The Effect of Warm Local Anesthetic Solution on Epidural Anesthesia
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Eun MI, Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: kangnamANE
Record Dates: First submitted 2019-01-25; First posted 2019-03-01 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Cesarean Section
Keywords: pre-warmed epiural anesthetics; epidural anesthesia
MeSH Terms: interventions — Temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-warmed drug: Pre-warmed (38°C) ropivacaine (7.5mg/ml) 19ml and fentanyl 50ug are injected via the epidural route at the L3-4 interspace.
  Interventions: Other: Temperature
- Room temperature drug: Room temperature (20°C) ropivacaine (7.5mg/ml) 19ml and fentanyl 50ug are injected via the epidural route at the L3-4 interspace.

INTERVENTIONS:
Other: Temperature — temperature of drug
  Groups: Pre-warmed drug

SUMMARY:
The investigators are going to compare the onset and duration of nerve blockage with the use of pre-warmed (38°C) and room temperature (20°C) local anesthetic solutions (ropivacaine and fentanyl) on epidural anesthesia for cesarean section, and compare the incidence of complications such as hypotension, nausea and vomiting.

DETAILED DESCRIPTION:
Spinal anesthesia has a shorter time to onset than epidural anesthesia, and the amount of local anesthetic administered is lower than that of epidural anesthesia, resulting in less systemic toxicity and superior block effect.

However, there are disadvantage that it is difficult to control the block height and the incidence of hypotension is high.

On the other hand, epidural anesthesia has the advantages of less sudden hypotension due to slow autonomic blockade, but it has a disadvantage that sensory nerve and motor nerve block time is delayed compared to spinal anesthesia.

The degree of nerve block for cesarean section surgery requires a high level of anesthesia above the T6 level, so the frequency of hypotension is high due to rapid sympathetic block after spinal anesthesia.

In this respect, hemodynamically stable epidural anesthesia is preferred when performing anesthesia for cesarean section.

The investigators are going to compare the onset and duration of nerve blockage with the use of pre-warmed (38°C) and room temperature (20°C) local anesthetic solutions (ropivacaine and fentanyl) on epidural anesthesia for cesarean section, and compare the incidence of complications such as hypotension, nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Among the pregnant women who were administered cesarean section in this study, those who agreed to participate in this study.

Exclusion Criteria:

* Fetal distress requiring fast delivery.
* Patients with hypersensitivity, allergic response, resistance to the drugs used in this study (fentanyl, ropivacaine, lidocaine).
* Patients who is not possible for regional anesthesia
* Patients who refused to participate in this study.
* Patients who cannot read or understand the agreement.
* Patients whose weight is less than 50kg or exceeds 100kg.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Among the pregnant women who were administered cesarean section in this study, those who agreed to participate in this study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Onset time of epidural anesthesia (up to T6 level) | During the operation
  After the administration of epidural local anesthetics the sensory block level is checked every 2 minutes for 20 minutes, every 10 minutes during operating period, and every 10 minutes for 60 minutes in the recovery room. The sensory block level is assessed using the pinprick test method.

SECONDARY OUTCOMES:
Incidence of hypotension | During the operation
  When systolic blood pressure is less than 90 mmHg or mean arterial pressure is less than 60 mmHg, 30 mcg of phenylephrine is administrated. If bradycardia(HR<50) is accompanied, 4mg of ephedrine is injected.
Incidence of nausea and vomiting | From the time of epidural injection to 1 hour after entering recovery room
  Record the nausea and vomiting that occurred in the operating room and in the recovery room after administration of the local anesthetic. If there is nausea and vomiting after surgery, ramosetron (0.3mg) should be administered if the postoperative nausea and vomiting(PONV) grade is 1 or more and symptoms are severe enough to require medication.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Mi Choi, MD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam sacred heart hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No